CLINICAL TRIAL: NCT02671994
Title: Significance of Geriatric Assessment for Optimal Treatment of Older Cancer Patients
Brief Title: Geriatric and Oncologic Assessment Before Treatment
Acronym: GOAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Sambavy Nadaraja, MD, PhD student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GOAT
Record Dates: First submitted 2016-01-27; First posted 2016-02-02 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Cancer
Keywords: Geriatric Assessment; G8 screening; Oncologic treatment
MeSH Terms: conditions — Neoplasms | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (experimental group) (Experimental): Oncologic treatment decision based on G8 screening followed by geriatric assessment and subsequent MDT, if needed, in addition to standard assessment (ECOG Performance Status + clinical assessment).
  Interventions: Other: G8 screening; Other: Geriatric assessment
- B (control group) (No Intervention): Oncologic treatment decision based on standard assessment (ECOG Performance Status + clinical assessment).

INTERVENTIONS:
Other: G8 screening
  Arms: A (experimental group)
Other: Geriatric assessment
  Arms: A (experimental group)

SUMMARY:
In a randomized controlled trial, the investigators wish to investigate, if oncologic treatment decision based on G8 screening followed by geriatric assessment and subsequent MDT, if needed, in older frail patients with gynaecologic and urologic cancer is superior to standard assessment (PS and clinical assessment) in oncologic treatment decision.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified gynaecologic cancer (ovarian, uterine, or cervical cancer) or urologic cancer (prostate, bladder, or kidney cancer).
* Suited for first line medical oncologic treatment with chemotherapy and/or targeted therapy.
* Age ≥ 70 years.
* Understands, speaks, and writes Danish.
* Signed informed consent.

Exclusion Criteria:

* Previous cancer diagnosis except for carcinoma in situ of the cervix or skin cancer other than malignant melanoma.
* Previous chemotherapy and/or targeted therapy for current cancer diagnosis.
* Previous radiation therapy or concomitant radiotherapy for current cancer diagnosis.
* Surgery within the last 4 weeks.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of planned oncologic treatment (number of participants, who complete the planned oncologic treatment) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jørn Herrstedt, MD, DMSc, Study Director — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nadaraja S, Matzen LE, Jorgensen TL, Dysager L, Knudsen AO, Jeppesen SS, Moller S, Herrstedt J; Academy of Geriatric Cancer Research (AgeCare). The impact of comprehensive geriatric assessment for optimal treatment of older patients with cancer: A randomized parallel-group clinical trial. J Geriatr Oncol. 2020 Apr;11(3):488-495. doi: 10.1016/j.jgo.2019.06.019. Epub 2019 Jul 3. PMID 31279749